CLINICAL TRIAL: NCT07121829
Title: A Phase 1b/2, Subprotocol of DAY101 in Combination With Pimasertib for Patients With Recurrent, Progressive, or Refractory Solid Tumors and MAPK Pathway Aberrations
Brief Title: Tovorafenib (DAY101) or in Combination With Pimasertib for Participants With Melanoma and Other Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Day One Biopharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAY101-102b; 2021-003768-29 (EudraCT Number)
Record Dates: First submitted 2025-07-03; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Melanoma; Solid Tumor; Pilocytic Astrocytoma; Non Small Cell Lung Cancer; Colorectal Cancer; Pancreatic Cancer; MAP Kinase Family Gene Mutation; RAS Mutation; RAF Mutation; MEK Mutation
Keywords: DAY101; Mitogen-activated protein kinase; tovorafenib; pimasertib; DAY201
MeSH Terms: conditions — Melanoma; Astrocytoma; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Pancreatic Neoplasms | interventions — tovorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Tovorafenib plus pimasertib
  Interventions: Drug: Tovorafenib; Drug: Tovorafenib Drug: Pimasertib

INTERVENTIONS:
Drug: Tovorafenib — Tovorafenib tablet for oral use.
Drug: Tovorafenib Drug: Pimasertib — Tovorafenib tablet for oral use. Pimasertib capsule for oral use

SUMMARY:
This is a subprotocol of Master Protocol DAY101-102 and is a Phase 1b/2, multi-center, open label subprotocol of participants ≥12 years of age, with recurrent or progressive solid tumors with alterations in the key proteins of the MAPK pathway, such as tumors that harbor RAS or RAF alterations.

*Note: Study concluded as Phase 1b only.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent by participant ≥12 years of age; either a Consent or an Assent Form will be provided to the patient based on their capacity, local regulations, and guidelines.
* Participants must have a report of histologically confirmed diagnosis of tumor and a concurrent MAPK pathway alteration (genomic alterations in RAS, RAF, MEK, or NF1) obtained through a tumor or liquid biopsy as assessed by genomic sequencing, polymerase chain reaction (PCR), fluorescence in situ hybridization (FISH), or another clinically accepted molecular diagnostic method recognized by local laboratory or regulatory agency
* Participants must have radiographically stable, recurrent or progressive disease that is measurable using the appropriate tumor response criteria eg, (RECIST version 1.1, RANO)
* Archival tumor tissue should be preferably less than 3 years old. If unavailable, a freshly acquired tumor tissue biopsy or liquid biopsy is required
* If brain metastases are present, they must have been previously treated and be stable as assessed by radiographic imaging

Exclusion Criteria:

* Known presence of concurrent activating alterations
* Participants with current evidence or a history of serous retinopathy (SR), retinal vein occlusion (RVO) or ophthalmopathy present at screening or baseline who would be considered at risk for SR or RVO
* Participants who have an unstable neurological condition, despite adequate treatment (eg, uncontrolled seizures)
* Participants with history of acute neurological events (such as intracranial or subarachnoid hemorrhage, stroke, intracranial trauma) within the past 6 months
* History of second malignancy within 3 years prior to study treatment except for curatively treated cervical cancer in situ, non-melanoma skin cancer, or superficial bladder cancer

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Number of participants who will report Treatment emergent adverse events (TEAEs) and serious TEAEs | Up to 30 days after the last dose of any study drug
Number of participants who will report clinically significant changes in vital signs | Up to 30 days after the last dose of any study drug
Number of participants who will report clinically significant changes in clinical chemistry parameters | Up to 30 days after the last dose of any study drug
Number of participants who will report clinically significant changes in hematology parameters | Up to 30 days after the last dose of any study drug
Number of participants with Dose limiting toxicities (DLTs) | Up to 30 days after the last dose of any study drug

SECONDARY OUTCOMES:
Percentage of participants with complete overall response rate (ORR) | Up to 30 months
  ORR as assessed by the proportion of participants with the best overall confirmed response of complete response (CR) or partial response (PR) according to the appropriate tumor response criteria as assessed by Investigator
Duration of response (DOR) | Up to 30 months
  The interval from the date of the first documentation of tumor response (CR or PR) that was subsequently confirmed by investigator assessment to the date of first occurrence of radiographic disease progression based on appropriate tumor response criteria as assessed by investigator or death due to any cause, whichever occurs earlier.
Progression Free Survival (PFS) | Up to 30 months
  The interval from the date of the first dose to the first occurrence of radiographic disease progression based on appropriate tumor response criteria as assessed by investigator or death due to any cause, whichever occurs earlier.
Overall Survival (OS) | Up to 30 months
  The interval from the date of the first dose until the recorded date of death due to any cause.
Time to Response | Up to 30 months
  Defined in participants with best overall response of CR or PR as determined by Investigator, time to response is defined as the interval from the date of the first dose to date of first documentation of tumor response (CR or PR) that was subsequently confirmed by investigator assessment.
Plasma concentration of DAY101 | Cycles 1 through Cycle 11 (each cycle is 28 days)
Maximum drug concentration (Cmax) of DAY101 | Cycle 1, Day 1 through Cycle 1, Day 22
Area Under the Curve from Time Zero to Last Measurable Concentration (AUC 0-last) | Cycle 1, Day 1 through Cycle 1, Day 22
Change in gene expression levels in pre and post treatment samples using RNA sequencing (RNA seq) analysis. | Up to 30 months
Change in expression levels of phosphorylated ERK (pERK) and Ki67 in pre and post treatment samples using immunohistochemistry methodology. | Up to 30 months

CONTACTS AND LOCATIONS:
Locations (10):
- United States (8):
  - The Angeles Clinic, Los Angeles, California
  - Hoag Health, Newport Beach, California
  - University of Colorado Hospital, Aurora, Colorado
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Community North Cancer Center, Indianapolis, Indiana
  - OHSU Knight Cancer Institute, Portland, Oregon
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - vanderbilt-Ingram Cancer Center, Nashville, Tennessee
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No